CLINICAL TRIAL: NCT02473354
Title: Predictors of Opioid-Induced Respiratory Depression (OIRD)
Acronym: (OIRD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00060429
Record Dates: First submitted 2015-06-03; First posted 2015-06-16 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Remifentanil; Oxygen; Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resp Depression Sequence 1 - 3 (Other): Sequence #1: breathe 21% through the facemask and increase ventilation to achieve a target hypocapnic ET CO2 of 25 - 30 mmHg. Subject will then breathe a gas mixture containing 6% CO2 / 30% O2 to achieve a target hypercapnic ET CO2 up to 60 mmHg or HCVR is terminated at the discretion of the PI.
  Sequence #2: breathe 21% O2 (normoxia) before remifentanil administration Sequence #3: breathe 50% O2 (hyperoxia) before remifentanil administration
  Interventions: Drug: Remifentanil; Drug: Oxygen; Drug: Carbon dioxide

INTERVENTIONS:
Drug: Remifentanil — The opioid used for this study is Remifentanil and is commonly used in the operating room. Remifentanil will be given under normoxic (breathing room air [21% Oxygen]) and hyperoxic (breathing 50% oxygen) conditions to determine if the measurement of the specific respiratory parameters will predict the OIRD response.
Drug: Oxygen — Remifentanil will be administered under normal oxygen (normoxia) and increased oxygen (hyperemic) conditions.
  Other Names: O2
Drug: Carbon dioxide — Carbon dioxide is used as part of the hypercapnia ventilatory response measurement (HCVR)
  Other Names: CO2

SUMMARY:
Purpose of the Study: (1) To classify an individual subject's ventilatory response in terms of respiratory depression to a bolus of remifentanil under normoxic and hyperoxic conditions. (2) Measurement of specific respiratory parameters to predict the opioid-induced respiratory depression (OIRD) response.

DETAILED DESCRIPTION:
This study is using FDA approved drugs (remifentanil, oxygen and carbon dioxide) in an investigational manner and the study is also developing a diagnostic test that is currently investigational. Investigational means that the FDA has not approved the use of the drugs in this manner or the diagnostic test being developed.

Opioid-Induced Respiratory Depression (OIRD) is recognized as potentially life threatening and the cause of substantial morbidity (poor health) and mortality (death). Respiratory depression is when the amount of breathing you do in a minute falls below normal. Opioids are medications widely used to treat both acute (lasting hours to days) and chronic (lasting months) pain, both within and outside the hospital setting. Opioids have been used outside the prescribed circumstances resulting in misuse and abuse. Even within the controlled environment of acute hospital care it is difficult to identify those individuals at most risk of OIRD, as many do not possess physical characteristics, such as obesity or obstructive sleep apnea (stop breathing during sleep), which may predispose to OIRD. In the absence of the ability to easily identify at-risk individuals the Anesthesia Patient Safety Foundation have suggested that all patients receiving opioids must be considered at risk of OIRD and therefore require appropriate monitoring.

Even when fully awake, the normal response to breathing a gas mixture containing carbon dioxide (CO2) is to increase the amount of breathing. The effect is similar to breathing in and out of a paper bag. This is called the Hypercapnic Ventilatory Response (HCVR) and can be measured. Not everyone responds in an identical manner - there will be differences in the HCVR from one person to the next. But if an individual's baseline HCVR is measured, then the change from baseline can also be measured.

This study is being done to: (1) classify or rate an individual subject's ventilatory (breathing) response in terms of respiratory depression to a bolus of a potent opioid (similar to morphine, often referred to as a narcotic). The opioid used for this study is Remifentanil and is commonly used in the operating room. Remifentanil will be given under normoxic (breathing room air [21% Oxygen]) and hyperoxic (breathing 50% oxygen) conditions to (2) determine if the measurement of the specific respiratory parameters will predict the OIRD response.

ELIGIBILITY:
Inclusion Criteria:

* is between 18 and 50 years of age;
* weighs greater than 40 kilograms;
* is American Society Anesthesiologist (ASA) status 1 [assessment by PI or delegate];
* has a BMI between 18.0 and 30.0 [calculated from measured height & weight];
* has completed the appropriate fasting periods for solids and liquids prior to the administration of remifentanil
* and has provided written informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* has a prior or known allergy to lidocaine or similar pharmacologic agents;
* is currently taking any medication other than for birth control;
* is currently participating in, or has recently participated in (discontinued within 30 days prior to this study) in an investigational drug study [self-reported];
* has a negative Allen's Test to confirm patency of the collateral artery [clinical assessment by PI or delegate];
* has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported];
* is female with a positive pregnancy test [serum or urine], or is female and is unwilling to use effective birth control between the time of screening and study procedure;
* has anemia [measured by venous blood gas sample];
* has a history of sickle cell disease [self-reported];
* has a positive urine cotinine or urine drug screen or oral ethanol test [POC testing];
* has a history of narcotic or recreational drug addition [self reported by subject in response to questioning by PI or delegate; review of duke electronic medical history record];
* has room air saturation less than 95% by pulse oximetry [measurement by PI or delegate];
* has a clinically significant abnormal EKG [assessment by PI or delegate];
* has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
* has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co-oximetry];
* is intolerant to a breathing mask apparatus [assessment by PI or delegate];
* has any condition in the opinion of the investigator which would make him or her unsuitable for study participation [assessment by PI or delegate];
* is unwilling or unable to provide informed consent or comply with the study procedures;
* has Rayanud's disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Hypercapnic Ventilatory Response (HCVR) gradient based upon ETCO2 and Minute Volume | Sequence #1 approximately 30 minutes
  Is there a correlation between the HCVR and susceptibility of OIRD.

SECONDARY OUTCOMES:
The proportion of subjects who are classified as low, medium, or high risk for Opioid Induced Respiratory Depression (OIRD). | Sequence #2 approximately 1 hour
  This will be measure in Low, Medium, or High.

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MB BS, Principal Investigator — Duke Anesthesiology
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided